CLINICAL TRIAL: NCT00805740
Title: Efficacy And Safety Of Eraxis/Ecalta (Anidulafungin) Compared To Cancidas (Caspofungin) In Patients With Candida Deep Tissue Infection
Brief Title: An Evaluation Of The Effectiveness And Safety Of Anidulafungin Compared To Caspofungin For The Treatment Of Deep Tissue Infection Due To Candida
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated prematurely on May 18, 2012 due to slow enrollment. The study was not terminated due to any safety issues or concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A8851022
Record Dates: First submitted 2008-11-26; First posted 2008-12-10 (Estimated); Results first posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-05

CONDITIONS: Candidiasis; Fungemia
Keywords: Candidiasis; Invasive Candidiasis; Deep Tissue Candidiasis; Candida; Candidemia; Fungal Infection
MeSH Terms: conditions — Candidiasis; Fungemia; Candidiasis, Invasive; Torulopsis; Candidemia; Mycoses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anidulafungin arm (Experimental)
  Interventions: Drug: Active anidulafungin
- Caspofungin arm (Experimental)
  Interventions: Drug: Active Caspofungin

INTERVENTIONS:
Drug: Active anidulafungin — Subjects in this arm will receive active anidulafungin and placebo caspofungin
  Arms: Anidulafungin arm
Drug: Active Caspofungin — Subjects in this arm will receive active caspofungin and placebo anidulafungin
  Arms: Caspofungin arm

SUMMARY:
The purpose of this study is to gather information on the use of anidulafungin for the treatment of serious Candida infection. It is expected that anidulafungin will be at least as safe and as effective as the comparator drug, caspofungin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of deep tissue Candida infection, defined as growth of Candida sp. from a culture specimen obtained from a normally sterile site accompanied by signs and symptoms of infection.
* Male or female ≥ 16 years of age.
* Expected hospitalization for at least fourteen (14) days.

Exclusion Criteria:

* Pregnancy or breast feeding or planning to become pregnant during the study.
* Recent treatment with one of the study drugs over the last 30 days.
* Allergy to either study drug or to this class of drugs.
* Significant liver dysfunction.
* Suspected Candida osteomyelitis, endocarditis, meningitis or any other infections of the central nervous system.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- United States (3):
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Wilmington, Delaware
  - Pfizer Investigational Site, Detroit, Michigan
- Belgium (2):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Brussels
- Pfizer Investigational Site, Sofia, Bulgaria
- Pfizer Investigational Site, Vancouver, British Columbia, Canada
- Netherlands (2):
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Nijmegen
- Portugal (2):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Lisbon
- Pfizer Investigational Site, Bucharest, Romania
- Pfizer Investigational Site, P/o Stepanovskoe, Krasnogorskiy District, Moscow Region, Russia
- Pfizer Investigational Site, Geneva, Switzerland

REFERENCES:
- [Derived] De Rosa FG, Busca A, Capparella MR, Yan JL, Aram JA. Invasive Candidiasis in Patients with Solid Tumors Treated with Anidulafungin: A Post Hoc Analysis of Efficacy and Safety of Six Pooled Studies. Clin Drug Investig. 2021 Jun;41(6):539-548. doi: 10.1007/s40261-021-01024-7. Epub 2021 Apr 23. PMID 33891293
- [Derived] Sganga G, Wang M, Capparella MR, Tawadrous M, Yan JL, Aram JA, Montravers P. Evaluation of anidulafungin in the treatment of intra-abdominal candidiasis: a pooled analysis of patient-level data from 5 prospective studies. Eur J Clin Microbiol Infect Dis. 2019 Oct;38(10):1849-1856. doi: 10.1007/s10096-019-03617-9. Epub 2019 Jul 6. PMID 31280481
- [Derived] Kontoyiannis DP, Bassetti M, Nucci M, Capparella MR, Yan JL, Aram J, Hogan PA. Anidulafungin for the treatment of candidaemia caused by Candida parapsilosis: Analysis of pooled data from six prospective clinical studies. Mycoses. 2017 Oct;60(10):663-667. doi: 10.1111/myc.12641. Epub 2017 Jun 9. PMID 28597967
- [Derived] Kullberg BJ, Vasquez J, Mootsikapun P, Nucci M, Paiva JA, Garbino J, Yan JL, Aram J, Capparella MR, Conte U, Schlamm H, Swanson R, Herbrecht R. Efficacy of anidulafungin in 539 patients with invasive candidiasis: a patient-level pooled analysis of six clinical trials. J Antimicrob Chemother. 2017 Aug 1;72(8):2368-2377. doi: 10.1093/jac/dkx116. PMID 28459966
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851022&StudyName=An%20Evaluation%20Of%20The%20Effectiveness%20And%20Safety%20Of%20Anidulafungin%20Compared%20To%20Caspofungin%20For%20The%20Treatment%20Of%20Deep%20Tissue%20Infection%20Due%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Anidulafungin: Anidulafungin at a loading dose 200 milligram (mg) as two 100 mg consecutive infusions intravenously over 1.5 hours each, administered prior to or following placebo matched to caspofungin 70 mg infusion intravenously over 1 hour on Day 1. Anidulafungin 100 mg infusion intravenously over 1.5 hours once daily, administered prior to or following placebo matched to caspofungin 50 mg infusion intravenously over 1 hour once daily starting from Day 2 to end of treatment (Day 14 to Day 42).
- Caspofungin: Caspofungin at a loading dose 70 mg infusion intravenously over 1 hour, administered prior to or following 2 placebo infusions, each matched to anidulafungin 100 mg infusion, intravenously over 1.5 hours each on Day 1. Caspofungin 50 mg infusion intravenously over 1 hour once daily, administered prior to or following placebo matched to anidulafungin 100 mg infusion intravenously over 1.5 hours once daily starting from Day 2 to end of treatment (Day 14 to Day 42).
Period: Overall Study
Arm/Group | Anidulafungin | Caspofungin
Started | 28 | 13
Treated | 26 | 13
Completed | 17 | 9
Not Completed | 11 | 4
Not completed — Death | 7 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Randomized, but not treated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anidulafungin | Caspofungin | Total
Number analyzed (Participants) | 26 | 13 | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 56.3 (16.2) | 63.4 (16.3) | 58.6 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 17 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Global Response at End of Treatment (Day 14 To Day 42)
Description: Participants had successful global response if there was clinical response of cure/improvement,microbiological eradication/presumed eradication.Clinical cure:resolution of signs/symptoms (s/s) of Candida infection;no additional systemic/oral antifungal treatment needed.Clinical improvement:significant,but incomplete resolution of s/s of Candida infection;no additional systemic/oral antifungal treatment needed.Microbiological eradication/presumed eradication:baseline pathogen not isolated from original site culture,or culture data not available for participant with successful clinical outcome.
Time Frame: End of Treatment (Day 14 to Day 42)
Population: Modified Intent-To-Treat (MITT) population included all participants who received at least 1 dose of study drug and had a positive culture for Candida species (sp.).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 24 | 13
percentage of participants | 83.3 [62.6 to 95.3] | 61.5 [31.6 to 86.1]
Statistical Analysis 1: Comparison: Anidulafungin vs Caspofungin; The 95 percent (%) confidence interval (CI) was calculated using method of exact unconditional confidence limits for the difference. Global response (rates of success) by using a 2-sided 95% CI for the true difference in efficacy (Anidulafungin minus Caspofungin) was calculated. Statistical testing was done at 2.5% alpha; Test type: Superiority or Other; Risk Difference (RD) = 21.8, 95% CI 2-sided [-12.3 to 53.3]

2. Secondary Outcome: Percentage of Participants With Global Response at 2-week and 6-week Follow-up Visit
Description: as for outcome 1
Time Frame: 2-week follow-up (2 weeks after end of treatment [EOT]), 6-week follow-up (6 weeks after EOT)
Population: MITT population included all participants who received at least 1 dose of study drug and had a positive culture for Candida species. Only participants who completed therapy or who had global response of failure at EOT were evaluable for 2- and 6-week follow-up analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 21 | 11
percentage of participants
  2-week follow-up | 76.2 [52.8 to 91.8] | 54.5 [23.4 to 83.3]
  6-week follow-up | 66.7 [43.0 to 85.4] | 54.5 [23.4 to 83.3]
Statistical Analysis 1: Comparison: Anidulafungin vs Caspofungin; 2-week follow-up: The 95% CI was calculated using method of exact unconditional confidence limits for the difference. Global response (rates of success) by using a 2-sided 95% CI for the true difference in efficacy (Anidulafungin minus Caspofungin) was calculated. Statistical testing was done at 2.5% alpha; Test type: Superiority or Other; Risk Difference (RD) = 21.6, 95% CI 2-sided [-13.6 to 55.6]
Statistical Analysis 2: Comparison: Anidulafungin vs Caspofungin; 6-week follow-up: The 95% CI was calculated using method of exact unconditional confidence limits for the difference. Global response (rates of success) by using a 2-sided 95% CI for the true difference in efficacy (Anidulafungin minus Caspofungin) was calculated. Statistical testing was done at 2.5% alpha; Test type: Superiority or Other; Risk Difference (RD) = 12.1, 95% CI 2-sided [-23.3 to 47.3]

3. Secondary Outcome: Percentage of Participants With Response Based on Clinical Cure and Microbiological Success
Description: A participant had a successful response if there was clinical response of cure and microbiological success (eradication or presumed eradication). Clinical response of cure: resolution of signs and symptoms attributed to Candida infection; no additional systemic or oral antifungal treatment required to complete the course of therapy. Microbiological eradication or presumed eradication: baseline pathogen not isolated from original site culture, or culture data not available for a participant with successful clinical outcome.
Time Frame: EOT (Day 14 to 42), 2-week follow-up (2 weeks after EOT), 6-week follow-up (6 weeks after EOT)
Population: MITT population. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Here, 'n' signifies those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 21 | 8
percentage of participants
  EOT (n=21,8) | 81.0 | 62.5
  2-week follow-up (n=16,6) | 87.5 | 100.0
  6-week follow-up (n=15,6) | 93.3 | 100.0

4. Secondary Outcome: Percentage of Participants With Clinical Response
Description: A participant had a successful clinical response if there was clinical response of cure or improvement. Clinical response of cure: resolution of signs and symptoms attributed to Candida infection; no additional systemic or oral antifungal treatment required to complete the course of therapy. Clinical response of improvement: significant, but incomplete resolution of signs and symptoms of Candida infection; no additional systemic or oral antifungal treatment required.
Time Frame: Day 10
Population: MITT population included all participants who received at least 1 dose of study drug and had a positive culture for Candida species.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 24 | 13
percentage of participants | 70.8 [48.9 to 87.4] | 76.9 [46.2 to 95.0]
Statistical Analysis 1: Comparison: Anidulafungin vs Caspofungin; The 95% CI was calculated using method of exact unconditional confidence limits for the difference. Global response (rates of success) by using a 2-sided 95% CI for the true difference in efficacy (Anidulafungin minus Caspofungin) was calculated. Statistical testing was done at 2.5% alpha; Test type: Superiority or Other; Risk Difference (RD) = -6.1, 95% CI 2-sided [-39.0 to 27.9]

5. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse was defined as any baseline Candida sp. isolated following eradication (documented or presumed) or culture data not available for participants with a clinical response of failure after a previous response of success. Prophylactic treatment with oral antifungal agents was not sufficient to document a relapse.
Time Frame: 2-week follow-up (2 weeks after EOT), 6-week follow-up (6 weeks after EOT)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 24 | 13
percentage of participants
  2-week follow-up | 0 | 0
  6-week follow-up | 0 | 0

6. Secondary Outcome: Percentage of Participants With New Infection
Description: New Infection: participant presenting with clinical failure with the emergence of new Candida sp. at the original site of infection or at a distant site of infection. Clinical failure: no significant improvement in signs and symptoms, or death due to Candida infection. Participants must have had received at least 3 doses of study drug to be classified as a failure.
Time Frame: 2-week follow-up (2 weeks after EOT), 6-week follow-up (6 weeks after EOT)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 24 | 13
percentage of participants
  2-week follow-up | 0 | 0
  6-week follow-up | 0 | 0

7. Secondary Outcome: Time to Negative Blood Culture
Description: Negative blood culture referred to absence of Candida sp. in the blood sample of participants who had a positive blood culture at baseline. Time to negative blood culture (days) was calculated as date of first negative blood culture minus first treatment date plus 1.
Time Frame: Baseline up to 6-week follow-up (6 weeks after EOT)
Population: A sub-set of MITT population included only those participants who had a positive blood culture for Candida species at baseline.
Measure: Median (Full Range); unit: days
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 3 | 4
days | 2.0 [2 to 7] | 3.5 [2 to 10]

8. Secondary Outcome: Percentage of Participants With All-cause Mortality
Description: All-cause mortality during study therapy and at follow-up visits reported as unique death at EOT, 2 week follow-up and 6 week follow-up.
Time Frame: Baseline to EOT (Day 14 to 42), After EOT to 2-week follow-up (2 weeks after EOT), After 2-week follow-up to 6-week follow-up (6 weeks after EOT)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 26 | 13
percentage of participants
  Baseline to EOT | 3.8 | 15.4
  After EOT to 2-week follow-up | 15.4 | 15.4
  After 2-week follow-up to 6-week follow-up | 7.7 | 0.0

9. Secondary Outcome: Time to Death
Description: Time to death (days) was assessed as date of death minus first treatment date plus 1.
Time Frame: Baseline up to 6-week follow-up (6 weeks after EOT)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: days
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 26 | 13
days | 23.0 [6 to 67] | 11.5 [9 to 51]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Anidulafungin | Caspofungin
Serious Adverse Events (participants affected / at risk) | 12/26 | 7/13
Other Adverse Events (participants affected / at risk) | 23/26 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin (N=26) | Caspofungin (N=13)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Injury associated with device (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Infectious peritonitis (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0
Nosocomial infection (Infections and infestations) | 1 | 0
Peptostreptococcus infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Splenic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin (N=26) | Caspofungin (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Coagulopathy (Blood and lymphatic system disorders) | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Eye disorder (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 1
Pupils unequal (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 1
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3
Chest pain (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Oedema (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Acinetobacter infection (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 1 | 0
Clostridium colitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Peritoneal candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Superinfection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Open wound (Injury, poisoning and procedural complications) | 1 | 0
Pancreatic leak (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Suture rupture (Injury, poisoning and procedural complications) | 1 | 0
Weaning failure (Injury, poisoning and procedural complications) | 1 | 0
Wound contamination (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Aspergillus test positive (Investigations) | 1 | 1
Bacterial test (Investigations) | 1 | 0
Bacterial test positive (Investigations) | 2 | 1
Bacteroides test positive (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 2
Blood bilirubin increased (Investigations) | 0 | 1
Blood culture negative (Investigations) | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 2
Blood triglycerides increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Citrobacter test positive (Investigations) | 0 | 1
Corynebacterium test positive (Investigations) | 0 | 1
Cytomegalovirus test positive (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Enterobacter test positive (Investigations) | 1 | 1
Enterococcus test positive (Investigations) | 0 | 2
Escherichia test positive (Investigations) | 0 | 2
Fungal test positive (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 1
Klebsiella test positive (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0
Platelet count increased (Investigations) | 0 | 1
Proteus test positive (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 1 | 0
Pseudomonas test positive (Investigations) | 1 | 0
Staphylococcus test positive (Investigations) | 1 | 3
Stenotrophomonas test positive (Investigations) | 1 | 0
Streptococcus test positive (Investigations) | 1 | 3
Urine output decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Catatonia (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Sleep disorder (Psychiatric disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urinoma (Renal and urinary disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Haemodynamic instability (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 2
Hypotension (Vascular disorders) | 3 | 3
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 2 | 2
Shock (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to slow enrollment. The study was not terminated due to any safety issues or concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.